CLINICAL TRIAL: NCT01398228
Title: Clinical Pathways for the Management of Acute Coronary Syndromes - Phase 3
Brief Title: Clinical Pathways for the Management of Acute Coronary Syndromes - Phase 3,CPACS-3
Acronym: CPACS-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Responsible Party: Principal Investigator, Yangfeng Wu, senior director, The George Institute for Global Health, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CPACS-3
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Acute Coronary Syndromes
Keywords: Quality of care; Acute Coronary Syndromes (ACS)
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Other): Group 1 will receive quality improvement initiatives first, after 6 months of baseline initiation.
  Interventions: Behavioral: quality improvement initiatives
- Group 2 (Other): Group 2 will receive quality improvement initiatives second, after 6 months of the intervention initiation for Group 1.
  Interventions: Behavioral: quality improvement initiatives
- Group 3 (Other): Group 3 will receive quality improvement initiatives third, after 6 months of the intervention initiation for Group 2.
  Interventions: Behavioral: quality improvement initiatives
- Group 4 (Other): Group 4 will receive quality improvement initiatives forth, after 6 months of the intervention initiation for Group 3.
  Interventions: Behavioral: quality improvement initiatives

INTERVENTIONS:
Behavioral: quality improvement initiatives — A six component quality improvement intervention will be implemented. These components include: establishment of a quality improvement team, hospital performance audit and feedback, implementation of a clinical pathway, training of physicians and nurses, online technical support and patient education.

SUMMARY:
The burden of chronic, non-communicable disease, of which cardiovascular disease comprises a significant component, has increased rapidly and substantially in China over recent years. Over the coming decades China is predicted to experience a 69% increase in acute coronary disease(ACS), amounting to nearly 8 million additional events. A recent randomized trial of more than 15,000 patients with acute coronary syndromes, the second phase of Clinical Pathway for acute coronary syndromes in China (CPACS-2) study, showed that a quality improvement initiative could improve aspects of hospital care, including the proportion of patients discharged on appropriate medication. The study also identified a number of barriers to improved care including out of pocket costs and administration systems. However, the study was not able to determine the impact on clinical outcomes or the cost-effectiveness of the intervention. The aim of the third phase of the Clinical Pathway for acute coronary syndromes in China (CPACS-3) study is to determine whether a complex intervention comprising a clinical pathway for ACS management in combination with a number of physician and patient-oriented education tools can improve the quality of care and health outcomes among ACS patient admitted to resource-limited (provincial) hospitals. The effectiveness of the intervention will be evaluated using a cluster randomized trial (stepped wedge design) of ACS patients admitted to 104 hospitals in China. The study will incorporate two additional components (1) a qualitative substudy to identify the barriers and enablers to improved care and (2) a study comparing the cost-effectiveness of the intervention compared to usual care, from the perspective of the health care provider. The study will be conducted in conjunction with the Chinese Ministry of Health and the Chinese Society of Cardiology. The findings from CPACS3 will be able to inform health policy-makers about the extent to which quality improvement initiatives can reduce the risk of death and disability among the millions of ACS patients admitted to hospitals in China each year.

ELIGIBILITY:
Inclusion Criteria:

* admitted to participating hospitals
* diagnosed as Acute Coronary Syndromes(ACS) at the time of death or discharge
* aged 18 years or older

Exclusion Criteria:

* death happened within 10 mins after arriving hospital
* ACS happened during hospitalization due to other health problem
* patients already registered in the database

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29934 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
incidence rate of in-hospital major adverse cardiovascular events (MACE) | from hospitaliztion to 1 week after discharge
  In-hospital major adverse cardiovascular events (MACE) comprising all-cause mortality, myocardial infarction or recurrent myocardial infarction and non-fatal stroke.The in-hospital mortality will include patients who deid during hospitalization, patients who gave up treatment and home and die within 1 week after returning home, and patients transfer to superior hospitals but die within one day.

SECONDARY OUTCOMES:
in-hospital all cause deaths | from hospitaliztion to 1 week after discharge
  The in-hospital mortality will include patients who deid during hospitalization, patients who gave up treatment and home and die within 1 week after returning home, and patients transfer to superior hospitals but die within one day.
a patient level composite score calculated by KPIs of ACS care | During Hospitalization, an expected average of 10 days
  A patient-level composite score is formed by dividing the total number of 15 pre-defined binary KPIs a patient receives by the total sum of KPIs a patient is eligible to receive. 15 KPI include: receive the first ECG within 10 minutes after arrival, receive aspirin within 24 hours of arrival, receive clopidogrel within 24 hours of arrival, receive statin within 24 hours of arrival, prescribe aspirin at discharge, prescribed clopidogrel at discharge, prescribed beta-blocker at discharge, prescribed statin at discharge, LVSD prescribed ACEI or ARB at discharge, STEMI that arrive hospital within 12 hours of symptom onset receive fibrinolysis, STEMI that received fibrinolytic therapy received this within 30 minutes of arrival, final diagnosis consistent with ECG and biomarker findings, receive both aspirin and clopidogrel within 24 hours, patient receive both aspirin and clopidogrel with loading dose within 24 hours, patient receive statin with loading dose within 24 hours.
each of the 16 KPIs (patient level) | During hospitalization, an expected average of 10 days
  receive the first ECG within 10 minutes after arrival, receive aspirin within 24 hours of arrival, receive clopidogrel within 24 hours of arrival, receive statin within 24 hours of arrival, prescribe aspirin at discharge, prescribed clopidogrel at discharge, prescribed beta-blocker at discharge, prescribed statin at discharge, LVSD prescribed ACEI or ARB at discharge, STEMI that arrive hospital within 12 hours of symptom onset receive fibrinolysis, STEMI that received fibrinolytic therapy received this within 30 minutes of arrival, final diagnosis consistent with ECG and biomarker findings, receive both aspirin and clopidogrel within 24 hours, patient receive both aspirin and clopidogrel with loading dose within 24 hours, patient receive statin with loading dose within 24 hours and length of stay.
a composite of MACE and re-hospitalization due to cardiovascular disease within 6 months after discharge | in 6 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yangfeng Wu, PhD, Principal Investigator — George Institute for global health, China
Locations (102):
- China (102):
  - Weining hospital, Bijie, Anhui
  - Lixin people's hospital, Bozhou, Anhui
  - Woyang people's hospital, Bozhou, Anhui
  - Wuwei people's hospital, Chaohu, Anhui
  - Yingshang people's hospital, Fuyang, Anhui
  - Linquan people's hospital, Fuyang, Anhui
  - Suixi people's hospital, Huaibei, Anhui
  - Shucheng people's hospital, Liuan, Anhui
  - Huoshang hospital, Liuan, Anhui
  - Zhuanglang people's hospital, Dingxi, Gansu
  - Gaolan people's hospital, Lanzhou, Gansu
  - Jingning people's hospital, Pingliang, Gansu
  - Zhuangliang people's hospital, Pingliang, Gansu
  - Taishan people's hospital, Jiangmen, Guangdong
  - Wuhua people's hospital, Meizhou, Guangdong
  - Lianzhou people's hospital, Qingyuan, Guangdong
  - Wuchuan people's hospital, Zhanjiang, Guangdong
  - Pu'an people's hospital, Buwei, Guizhou
  - Dejiang, Tongren, Guizhou
  - Yuqing people's hospital, Zunyi, Guizhou
  - Gaoyang hospital, Baoding, Hebei
  - Tang county hospital, Baoding, Hebei
  - Yi county hospital, Baoding, Hebei
  - Weichang manchu mongolia atounomous county hospital, Chengde, Hebei
  - Quzhou hospital, Handan, Hebei
  - Jizhou hospital, Jizhou, Hebei
  - Qinglong hospital, Qinhuangdao, Hebei
  - Zanhuang hospital, Shijiazhuang, Hebei
  - Shenze hospital, Shijiazhuang, Hebei
  - Pingxiang people's hospital, Xingtai, Hebei
  - Huaxian people's hospital, Anyang, Henan
  - Wuzhi people's hospital, Jiaozuo, Henan
  - Ruyang people's hospital, Luoyang, Henan
  - Xixia people's hospital, Nanyang, Henan
  - Chang huan hong li hospital, Xinxiang, Henan
  - Shangcheng people's hospital, Xinyang, Henan
  - Dancheng people's hospital, Zhoukou, Henan
  - Pingyu people's hospital, Zhumadian, Henan
  - Jianshi people's hospital, Enshi, Hubei
  - Songzi people's hospital, Jinzhou, Hubei
  - Danjiangkou's first hospital, Shiyan, Hubei
  - Tongcheng people's hospital, Xian'ning, Hubei
  - Gucheng people's hospital, Xiangfan, Hubei
  - Yidu's first hospital, Yichang, Hubei
  - Yingcheng people's hospital, Yingcheng, Hubei
  - Zhongxiang people's hospital, Zhongxiang, Hubei
  - Ba lin zuo qi people's hospital, Chifeng, Inner Mongolia
  - A rong qi people's hospital, Hulin, Inner Mongolia
  - Zha lu te people's hospital, Tongliao, Inner Mongolia
  - Huolinguole hospital, Tongliao, Inner Mongolia
  - DongHai people's hospital, Lianyungang, Jiangsu
  - Dongtai people's hospital, Yancheng, Jiangsu
  - Gaoyou people's hospital, Yangzhou, Jiangsu
  - Tongyu people's hospital, Baicheng, Jilin
  - Linjiang hospital, Baishan, Jilin
  - Dong feng people's hospital, Liaoyuan, Jilin
  - Qian'an hospital, Songyuan, Jilin
  - Huinan people's hospital, Tonghua, Jilin
  - Changbai montain protection and development zone central hospital, Yanbian, Jilin
  - Hunchun people's hospital, Yanbian, Jilin
  - Yitong 1st people's hospital, Yitong, Jilin
  - Beipiao 1st people's hospital, Chaoyang, Liaoning
  - Lingyuan people's hospital, Chaoyang, Liaoning
  - Zhuanghe central hospital, Dalian, Liaoning
  - Wafangdian people's hospital, Dalian, Liaoning
  - Kuandian Manchu Autonomous County Central Hospital, Dandong, Liaoning
  - Qingyuan Manchu Autonomous County people's hospital, Fushun, Liaoning
  - Beizhen people's hospital, Jinzhou, Liaoning
  - Changtu people's hospital, Tieling, Liaoning
  - Fengxiang hospital, Baoji, Shaanxi
  - Xixiang hospital, Hanzhong, Shaanxi
  - Mian county hospital, Hanzhong, Shaanxi
  - Fuping hospital, Weinan, Shaanxi
  - Hancheng people's hospital, Weinan, Shaanxi
  - Hu county hospital, Xi'an, Shaanxi
  - Zichang hospital, Yan’an, Shaanxi
  - Shenmu hospital, Yulin, Shaanxi
  - Chengwu people's hospital, Heze, Shandong
  - Pingyin people's hospital, Jinan, Shandong
  - Dong'e people's hospital, Liaocheng, Shandong
  - Yinan people's hospital, Linyi, Shandong
  - Xintai people's hospital, Tai’an, Shandong
  - Linqu people's hospital, Weifang, Shandong
  - Penglai people's hospital, Yantai, Shandong
  - Huantai people's hospital, Zibo, Shandong
  - Changzhi steel and iron group head hospital, Changzhi, Shanxi
  - Qingyuan people's hospital, Changzhi, Shanxi
  - Hunyuan people's hospital, Datong, Shanxi
  - Gaoping people's hospital, Jincheng, Shanxi
  - Lingshi people's hospital, Jinzhong, Shanxi
  - Pu xian people's hospital, Linfen, Shanxi
  - Xiangfen people's hospital, Linfen, Shanxi
  - Guxian people's hospital, Linfen, Shanxi
  - Yicheng people's hospital, Linfen, Shanxi
  - Lou fan people's hospital, Taiyuan, Shanxi
  - Houma people's hospital, Xintian, Shanxi
  - Yuanping people's hospital, Xinzhou, Shanxi
  - Huanqu people's hospital, Yuncheng, Shanxi
  - Dazhu people's hospital, Dazhou, Sichuan
  - Cangxi people's hospital, Guangyuan, Sichuan
  - Mianning people's hospital, Liangshan, Sichuan
  - Xuyong people's hospital, Luzhou, Sichuan

REFERENCES:
- [Derived] Xie G, Patel A, Du X, Sun Y, Li X, Wu T, Hao Z, Gao R, Wu Y. Impact of In-Hospital Quality of Care Improvement Initiative on Secondary Prevention of Acute Coronary Syndrome in Six Months After Patient Discharge: A Large Stepped Wedge- and Cluster-Randomized Controlled Trial. Circ Cardiovasc Qual Outcomes. 2025 May;18(5):e011441. doi: 10.1161/CIRCOUTCOMES.124.011441. Epub 2025 Apr 4. PMID 40184150
- [Derived] Xie W, Patel A, Boersma E, Feng L, Li M, Gao R, Wu Y. Chronic kidney disease and the outcomes of fibrinolysis for ST-segment elevation myocardial infarction: A real-world study. PLoS One. 2021 Jan 19;16(1):e0245576. doi: 10.1371/journal.pone.0245576. eCollection 2021. PMID 33465135
- [Derived] Sun Y, Feng L, Li X, Gao R, Wu Y. The sex difference in 6-month MACEs and its explaining variables in acute myocardial infarction survivors: Data from CPACS-3 study. Int J Cardiol. 2020 Jul 15;311:1-6. doi: 10.1016/j.ijcard.2020.03.043. Epub 2020 Mar 20. PMID 32223960
- [Derived] Feng L, Li M, Xie W, Zhang A, Lei L, Li X, Gao R, Wu Y. Prehospital and in-hospital delays to care and associated factors in patients with STEMI: an observational study in 101 non-PCI hospitals in China. BMJ Open. 2019 Nov 10;9(11):e031918. doi: 10.1136/bmjopen-2019-031918. PMID 31712344
- [Derived] Wu Y, Li S, Patel A, Li X, Du X, Wu T, Zhao Y, Feng L, Billot L, Peterson ED, Woodward M, Kong L, Huo Y, Hu D, Chalkidou K, Gao R; CPACS-3 Investigators. Effect of a Quality of Care Improvement Initiative in Patients With Acute Coronary Syndrome in Resource-Constrained Hospitals in China: A Randomized Clinical Trial. JAMA Cardiol. 2019 May 1;4(5):418-427. doi: 10.1001/jamacardio.2019.0897. PMID 30994898
- [Derived] Li S, Wu Y, Du X, Li X, Patel A, Peterson ED, Turnbull F, Lo S, Billot L, Laba T, Gao R; CPACS-3 investigators. Rational and design of a stepped-wedge cluster randomized trial evaluating quality improvement initiative for reducing cardiovascular events among patients with acute coronary syndromes in resource-constrained hospitals in China. Am Heart J. 2015 Mar;169(3):349-55. doi: 10.1016/j.ahj.2014.12.005. Epub 2014 Dec 18. PMID 25728724